CLINICAL TRIAL: NCT02802943
Title: iVAC-CLL01: Patient-individualized Peptide Vaccination After First Line Therapy of CLL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Robert Bosch Gesellschaft für Medizinische Forschung mbH (RBMF) (Other); Klinikum Stuttgart (Other); Marienhospital Stuttgart (Other); Katharinenhospital Stuttgart (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: iVAC-CLL01:
Record Dates: First submitted 2016-03-23; First posted 2016-06-16 (Estimated); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Leukemia, Chronic Lymphatic
Keywords: CLL, Peptid Vaccination
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Protein Subunit Vaccines; Imiquimod

STUDY DESIGN:
Intervention Model Description: MRD-negative (MRD-) patients (flow cytometry based, CLL cells in peripheral blood and bone marrow <10-4 6-10 weeks after the end of first line treatment).
  MRD-positive (MRD+) patients (flow cytometry based, CLL cells in peripheral blood or bone marrow ≥ 10-4 6-10 weeks after the end of first line treatment)
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peptide Vaccine MRD + (Experimental): MRD-positive (MRD+) patients (flow cytometry based, CLL cells in peripheral blood or bone marrow ≥ 10-4 6-10 weeks after the end of first line treatment)
  Interventions: Biological: Peptide Vaccine; Drug: Imiquimod
- Peptide Vaccine MRD- (Experimental): MRD-negative (MRD-) patients (flow cytometry based, CLL cells in peripheral blood and bone marrow <10-4 6-10 weeks after the end of first line treatment)
  Interventions: Biological: Peptide Vaccine; Drug: Imiquimod

INTERVENTIONS:
Biological: Peptide Vaccine — Individualized multi-peptide cocktail consisting of 300 μg each of 5 HLA class I and 4 HLA class II restricted peptides. The peptides for each individual patient will be selected from a warehouse consisting of 30 different peptides restricted by the 6 most common HLA class I allotypes (A*01, A*02, A*03, A*24, B*07, B*08) and 4 HLA class II peptides. Peptides will be administered subcutaneously. Vaccination will take place on d1, d4, d8, d15, d22 followed by vaccinations every 4 weeks for 1 year. The peptide warehouse is selected based on our data on the non-mutant HLA-presented antigenome of CLL identified as frequently presented CLL-associated T cell epitopes with a high potential for broad clinical application.
Drug: Imiquimod — All patients will receive imiquimod (Aldara®) as local adjuvant, applied topically at the side of vaccination 18h to 24h prior to the vaccination.

SUMMARY:
The aim of this study is to induce a peptide-specific immune response in CLL patients by multi-peptide vaccination with a patient-individualized peptide cocktail.

DETAILED DESCRIPTION:
Study Duration and Schedule:

The duration of the trial for each subject is expected to be 24 months. The duration for each individual patient includes about 6 months first-line therapy according to treating physicians choice with HLA ligandome analyses of CLL cells and selection of patient-individual multipeptide vaccine being performed in parallel, 12 months study treatment and 6 months followup time. The overall duration of the trial is expected to be approximately 4 years. Recruitment of subjects will start in 09/2016. The actual overall duration or recruitment may vary.

General Criteria for Subject Selection:

For the screening procedures of this study, physically fit subjects (as defined by ECOG score ≤2) with a confirmed diagnosis of a CLL/SLL according to the IWCLL guidelines requiring treatment are eligible. First line treatment will be performed according to treating physicians choice. The trial population will consist of both genders. Gender distribution in the trial is supposed to reflect the distribution in the real patient's population (approx. 60% male and 40% female patients), i.e. there will be no prior defined quantitative ratio between females and males. To assure that the included patients have the ability to mount an immune response, immune response to an HLA matched EBV/CMV peptide mix will be assessed in the screening phase. 60ml blood will be taken at the screening study visit. Peripheral mononuclear cells will be isolated and analyzed in a 12 day IFNγ ELISPOT for memory Tcell response to an EBV/CMV peptide mix. Only patients showing a positive immune response (section 8.1.1) will be eligible to receive the study drugs after first line treatment.

For the study treatment, physically fit subjects (as defined by ECOG score ≤2) with a confirmed diagnosis of CLL according to the IWCLL guidelines, which were treated with a first line therapy according to physicians choice are eligible. Subjects must have achieved at least a PR (IWCLL guidelines for the diagnosis and treatment of CLL) after treatment with first line therapy.The end of study is determined as the date of the last visit of the last patient (LSO 04/2020).

Study Design:

Interventional, open-label, multi-center phase II trial with use of a patient-individualized multipeptide vaccine and imiquimod as adjuvant

Blinding:

No blinding will be performed to avoid unnecessary complications of intradermal injections with sodium acid solution. Method against bias in patient selection: The patient selection will be documented. Reasons for refusal will be assessed.Method against bias in treatment manualized treatment protocol, monitoring and treatment reports. Method against bias in data analysis: Monitoring, analysis by intention to treat; independent statistician.

Chronic lymphatic leukaemia-peptide vaccine (CLL-VAC) drug product (DP):

Each patient enrolled in the iVAC-CLL01 trial will receive a CLL-VAC DP specifically tailored to the individual HLA ligandome of his/her respective CLL cells. The DPs are composed of peptides that are first manufactured as drug substances. A process named CLL-VAC_v1 enables the selection of drug substances to compose the unique, patient individual CLL-VAC DPs. CLL-VAC DPs will be composed based on a peptide warehouse consisting of 40 individual peptides (drug substances; 30 HLA class I peptides (5 A*01, 5 A*02, 5 A*03, 5 A*24, 5 B*07, 5 B*08) and 4 HLA class II peptides. All HLA class I peptides and HLA class II peptides are shown to be immunogenic. For each patient 5 HLA class I peptides are selected from the warehouse based on patient individual HLA ligandome analysis of CLL cells and are subsequently formulated into the personalized drug; the 4 HLA class II peptides will be included in each peptide vaccine cocktail.

All warehouse peptides are manufactured by BCN PEPTIDES, S.A, Els Vinyets-Els Fogars II, 08777 Sant Quintí de Mediona (Barcelona), Spain, or by Wirkstoffpeptidlabor, University of Tübingen, Auf der Morgenstelle 15, 72076 Tübingen, Germany. Both production sites hold certificates for the production of GMP grade synthetic peptides. All peptides are synthetic peptides, which will be manufactured by well-established solid phase peptide synthesis (SPPS) procedures using Fmoc chemistry.

Aldara® (imiquimod) Cream, 5%, is supplied as in single-use packets (24 per box), each of which contains 250 mg of the cream, equivalent to 12.5 mg of imiquimod. Aldara® (Meda GmbH) is a standard good of release.

ELIGIBILITY:
1. Documented diagnosis of CLL/SLL according to IWCLL guidelines.

   For Screening phase:
   * No pretreatment of CLL/SLL
   * Ability to mount an immune response: Positive immunresponse to EBV/CMV peptide mix (analyzed in 12 day recall IFNγ ELISPOT).

   For Vaccination phase:

   • Achievement of response (at least PR according to IWCLL guidelines) after first-line therapy according to treating physicians choice.
2. HLA typing positive for HLA alleles of peptides included in the warehouse with proven immunogenicity: HLA-A*01, A*02, A*03, A*24, B*07, B*08.
3. Ability to understand and voluntarily sign an informed consent form.
4. Age ≥ 18 years at the time of signing the informed consent form.
5. Ability to adhere to the study visit schedule and other protocol requirements.
6. Eastern Cooperative Oncology Group (ECOG) performance status score of ≤ 2.
7. Negative serological Hepatitis B and C test or negative PCR in case of positive serological test without evidence of an active infection, negative HIV test within 6 weeks prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2016-10-05 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-11-18 (Actual)

PRIMARY OUTCOMES:
Induction of peptide-specific T cell responses | 6 month after start of therapy
  The rate of patients with induction of peptide-specific T cell responses within a maximum of 6 month after start of therapy will be the primary endpoint for efficacy.
  Analysis of the primary endpoint= induction of immune response:
  The induction of peptide-specific T cell responses will be determined by IFNγ ELISPOT.
  T cell responses will be considered to be positive when >15 spots/well (IFNγ ELISPOT) were counted and the mean spot count per well is at least 3-fold higher than the mean number of spots in the negative control wells (according to the cancer immunoguiding program guidelines).

SECONDARY OUTCOMES:
Overall Survival | 6 month after start of therapy
  Secondary endpoints will be the overall survival, the disease free survival and the remission status at the end of study, the achievement of MRD-negativity or reduction in MRD-positive patients as well as safety and toxicity (CTCAE V 4.03)

CONTACTS AND LOCATIONS:
Locations (5):
- Germany (5):
  - Katharinenhospital, Stuttgart, Baden-Wurttemberg
  - Diakonie-Klinikum Stuttagrt, Stuttgart, Baden-Wurttemberg
  - Marienhospital, Stuttgart, Baden-Wurttemberg
  - Robert-Bosch-Krankenhaus Abteilung fuer Haematologie, Onkologie und Palliativmedizin, Stuttgart, Baden-Wurttemberg
  - University Hospital Tuebingen, Tübingen, Baden-Wurttemberg

REFERENCES:
- [Derived] Heitmann JS, Jung S, Wacker M, Maringer Y, Nelde A, Bauer J, Denk M, Hoenisch-Gravel N, Richter M, Oezbek MT, Dubbelaar ML, Bilich T, Pumptow M, Martus P, Illerhaus G, Denzlinger C, Steinbach F, Aulitzky WE, Muller MR, Dorfel D, Rammensee HG, Salih HR, Walz JS. Warehouse-based, immunopeptidome-guided design of personalised peptide vaccines shows feasibility in clinical trial evaluation in CLL patients. Front Immunol. 2024 Nov 26;15:1482715. doi: 10.3389/fimmu.2024.1482715. eCollection 2024. PMID 39660140